CLINICAL TRIAL: NCT05745805
Title: Cohort Follow-up of Epidemic and Neuroimaging for Patients During the 1st Wave of the COVID-19 in China
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Nuclear 215 Hospital of Shaanxi Province (Unknown); Yanan Traditional Chinese Medicine Hospital (Unknown); Shangluo Central Hospital (Other); Xian QinHuang Hospital (Unknown); Yulin No.2 Hospital (Other); Hanzhong Central Hospital (Other); Ankang Central Hospital (Other); Baoji High-tech Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2023-012
Record Dates: First submitted 2023-02-24; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: COVID-19; Post-COVID-19 Syndrome; Acute COVID-19; Post-Acute COVID-19
Keywords: COVID-19; Post-COVID-19 Syndrome; Neuroimaging; Epidemic; Simultaneous Cortico-Spinal Magnetic Resonance Imaging
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild COVID-19 group: Confirmed diagnosis of mild Covid-19 (WHO criteria)
  Interventions: Device: Simultaneous cortico-spinal magnetic resonance imaging, Serum
- Moderate COVID-19 group: Confirmed diagnosis of moderate Covid-19 (WHO criteria)
  Interventions: Device: Simultaneous cortico-spinal magnetic resonance imaging, Serum
- Uninfected Healthy controls: Healthy people who have not had COVID-19
  Interventions: Device: Simultaneous cortico-spinal magnetic resonance imaging, Serum

INTERVENTIONS:
Device: Simultaneous cortico-spinal magnetic resonance imaging, Serum — Simultaneous cortico-spinal magnetic resonance imaging data were collected in a strong magnetic field and collected the serum of participants.

SUMMARY:
Our main objective is to analyze the development of physical impact, mental health and blood profile over follow-up time during the 1st wave of the COVID-19. Besides, we aim to establish a database of post-COVID-19 based on simultaneous cortico-spinal magnetic resonance imaging data to identify high-risk patients with long COVID and prevent the neurological symptoms evolution, optimize the tactics of management in China.

DETAILED DESCRIPTION:
This is an observational, cross-sectional, and multicenter study. It will be performed at 9 public hospitals. Participants with confirmed cases of mild or moderate COVID-19 infection will complete the following programs at acute infection phase and after 3, 12 months for exploring biological mechanism and predictive biomarkers of post-COVID-19: 1) fill in the behavioral psychology scales, 2) submit blood samples at a local laboratory, 3) accept the simultaneous cortico-spinal magnetic resonance imaging scan. The uninfected healthy controls will complete the same programs as infected group mentioned above only at the time of inclusion. We will establish the simultaneous cortico-spinal magnetic resonance imaging database containing neuropsychological scales and blood parameters of post-COVID-19 in China.

ELIGIBILITY:
Inclusion Criteria:

Confirmed diagnosis of mild Covid-19 (WHO criteria)/Confirmed diagnosis of moderate Covid-19 (WHO criteria)/Healthy people who have not had COVID-19

Exclusion Criteria:

History of central nervous system diseases, such as mental disorder, degenerative diseases of central nervous system, tumors, trauma, etc. Participants with indication for MRI studies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be carried out in 9 hospitals among health team workers (doctors, nurses, employes) and social networks for patients who had a history of coronavirus infection COVID-19 confirmed by PCR analysis and antigen testing.
  The uninfected control population will be searched in the primary care services, media and social networks.
  All participants will sign informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2026-06-12 (Estimated); Study Completion 2026-09-12 (Estimated)

PRIMARY OUTCOMES:
Change in brain structure. | baseline and 3, 12 months
  The changes of brain volume (mm3) are evaluated by structural MRI
Change in brain function. | baseline and 3, 12 months
  The changes of brain functional connectivity intensity are evaluated by functional MRI

SECONDARY OUTCOMES:
Changes in symptoms assessed with a Symptom Checklist-90 Somatization (SCL-90 SOM) subscale. | baseline and 3, 12 months
  The 28 symptoms which are considered to be related to COVID-19 (headache, dizziness, chest pain, back pain, nausea, painful muscles, difficulties with breathing, feeling hot and cold alternately, tingling extremities, lump in the throat, general tiredness, heavy arms or legs, pain when breathing, runny nose, sore throat, dry cough, wet cough, fever, diarrhea, stomach pain, ageusia or anosmia, sneezing, and itchy eyes, fatigue, chest discomfort, tinnitus, anorexia and hypothermia) are assessed in participants with COVID-19. All symptoms are assessed using an ordinal 5-point Likert scale that answered to what extent participants were bothered by the respective symptom (1=not at all, 5=extremely) in the past 7 days.
Change in Fatigue. | baseline and 3, 12 months
  Fatigue is assessed with the Fatigue Impact Scale (FIS), Multidimensional Fatigue Inventory (MFI) and Fatigue Assessment Scale (FAS). A higher score represents a worse outcome.
  The FIS is a 40-item instrument assessing fatigue in three domains of daily life. Each item is rated on a five-step Likert scale, where 0 = no problems to 4 = extreme problems.
  The MFI is a 20-item self-report instrument covering four dimensions (general fatigue, physical fatigue, mental fatigue, reduced motivation and reduced activity) designed to measure fatigue.
  The FAS is an unidimensional fatigue scale and consisted of 10 items. The 5-point rating scale varies from 1, never, to 5, always.
Change in Post-Traumatic Stress Disorder. | baseline and 3, 12 months
  The PTSD is measured with the Impact of Events Scale-Revised (IES-R), a 22-item questionnaire designed to assess the participant's catastrophic experience of a particular life event. The 5-point rating scale varies from 0, not at all, to 4, extremely. A higher score corresponding to a worse outcome.
Change in pain. | baseline and 3, 12 months
  The pain intensity is assessed with the pain visual analogue scale (P-VAS). The The pain intensity varies from 0, no pain, to 10, Unbearable pain. A higher scores indicate greater pain intensity.
Change in cognition. | baseline and 3, 12 months
  The cognition is assessed with Montreal Cognitive Assessment (MoCA). Higher scores (0-30) are related to a better performance.
Change in executive function. | baseline and 3, 12 months
  The executive function is assessed with Trail Making Test A and B. Participants are asked to connect sequential numbers (TMT-A) and interconnect sequential numbers and letters (TMT-B).
Change in anxiety. | baseline and 3, 12 months
  Anxiety is assessed with Beck Anxiety Inventory (BAI). A higher score corresponding to more severe anxiety symptoms.
Change in Sleep. | baseline and 3, 12 months
  Sleep quality is assessed with Pittsburgh Sleep Quality Index (PSQI). A higher score corresponding to a worse sleep quality.
Change in depression. | baseline and 3, 12 months
  Depression is assessed with the Patient Health Questionnaire-9 (PHQ-9) and Beck Depression Inventory (BDI). A higher score corresponding to more severe depression symptoms.
Change in verbal memory. | baseline and 3, 12 months
  Verbal memory is assessed with the Auditory Verbal Learning Test (AVLT). A 12-word list are read by examiner three times and participants are asked to recall them followed by each presentation, which was called "immediate recall". The "short delayed recall" and "long delayed recall" ask the participants to recall the above 12-word list 5 minutes and 20 minutes later, the correctly recalled number of words are recorded. Finally, the subjects are instructed to recognize the learned words from a 24-words list which consisted of above learned 12-words list and a new unlearned 12-words list.
Change in working memory. | baseline and 3, 12 months
  Working memory is assessed with the Digit Span Backward. Participants are asked to repeat the numbers in the reverse order the examiner read them aloud and a higher score corresponding to a better outcome.
Change in auditory attention. | baseline and 3, 12 months
  Auditory attention is assessed with the Digit Span Forward. Participants are asked to repeat the numbers in the order the examiner read them aloud and a higher score corresponding to a better outcome.
Change in Inflammatory markers. | baseline and 3, 12 months
  The participants donate blood samples and the inflammatory markers will be analyzed with enzyme-linked immunosorbent assay (ELISA) Kit.
Change in Ig G and Ig M. | baseline and 3, 12 months
  The participants donate blood samples and the Ig G, Ig M will be analyzed with enzyme-linked immunosorbent assay (ELISA) Kit.
Change in myocardial enzymes. | baseline and 3, 12 months
  The participants donate blood samples and the creatine phosphokinase and lactic dehydrogenase will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhang, PhD, Principal Investigator — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Wu S, Luo Z, Liu H, Zhu J, Zhu Y, Hou D, Wei T, Liu T, Zheng C, Zhu Z, Huang W, Bai W, Yu X, Yuan H, Bao W, Zhang M, Niu X. Multicentre, multitime, multidimension, prospective follow-up cohort study on patients during the first wave of COVID-19 in China: a study protocol. BMJ Open. 2025 Jan 22;15(1):e083023. doi: 10.1136/bmjopen-2023-083023. PMID 39843379